CLINICAL TRIAL: NCT07312487
Title: Incidence, Associated Factors, and Management of Inadequate Analgesia During Cesarean Section Under Spinal Anesthesia in the Maternity Wards of the Strasbourg University Hospital: a 2-year Retrospective Study
Brief Title: Inadequate Analgesia During Cesarean Section Under Spinal Anesthesia
Acronym: ALGOCESA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9379
Record Dates: First submitted 2025-12-09; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Analgesia, Cesarean
Keywords: Analgesia During Cesarean; Spinal Anesthesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inadequate analgesia during cesarean section is a common condition, notably addressed by national recommendations from the SFAR (French Society of Anesthesia and Intensive Care) in 2021.

The objective of this study is to identify the specific characteristics of this condition in Strasbourg in terms of risk factors and management, and then to propose a protocol for its prevention and management.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman (age ≥18 years)
* Giving birth by cesarean section between January 1, 2021, and December 31, 2022, at the Strasbourg University Hospital

Exclusion Criteria:

* Patient who has expressed her opposition to the reuse of her data for scientific research purposes.

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: Adult woman (age ≥18 years) giving birth by cesarean section between January 1, 2021, and December 31, 2022, at the Strasbourg University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 2450 (Estimated)
Dates: Start 2024-10-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
General anesthesia rates | at day 1 post-operative

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésie Réanimation médecine Péri-Opératoire - Hôpitaux Universitaires de Strasbourg, Strasbourg, France